CLINICAL TRIAL: NCT00006305
Title: Bypass Angioplasty Revascularization Investigation in Type 2 Diabetes
Acronym: BARI2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maria Mori Brooks, Associate Professor of Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 133; U01HL061744 (NIH); U01HL061746 (NIH); U01HL061748 (NIH); U01HL063804 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Results first posted 2011-05-12 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases; Insulin Resistance; Diabetes Mellitus; Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases; Insulin Resistance; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Angioplasty; Coronary Artery Bypass; Biguanides; Thiazolidinediones; Insulin; Sulfonylurea Compounds; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Adrenergic beta-Antagonists; Calcium Channel Blockers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Revascularization and Insulin Providing (IP) (Active Comparator): Prompt revascularization with intensive medical therapy and insulin providing glycemic control strategy
  Interventions: Procedure: Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions; Procedure: Coronary Artery Bypass; Drug: Insulin, sulfonylurea; Drug: ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers
- Revascularization and Insulin Sensitizing (IS) (Active Comparator): Prompt revascularization with intensive medical therapy and insulin sensitizing glycemic control strategy
  Interventions: Procedure: Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions; Procedure: Coronary Artery Bypass; Drug: Biguanides, thiazolidinediones; Drug: ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers
- Medical Therapy and Insulin Providing (IP) (Active Comparator): Intensive medical therapy with delayed revascularization if clinically indicated and insulin providing glycemic control strategy
  Interventions: Drug: Insulin, sulfonylurea; Drug: ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers
- Medical Therapy and Insulin Sensitizing (IS) (Active Comparator): Intensive medical therapy with delayed revascularization if clinically indicated and insulin sensitizing glycemic control strategy
  Interventions: Drug: Biguanides, thiazolidinediones; Drug: ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers

INTERVENTIONS:
Procedure: Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions — Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions
  Arms: Revascularization and Insulin Providing (IP); Revascularization and Insulin Sensitizing (IS)
Procedure: Coronary Artery Bypass — Coronary Artery Bypass
  Arms: Revascularization and Insulin Providing (IP); Revascularization and Insulin Sensitizing (IS)
Drug: Biguanides, thiazolidinediones — Biguanides, thiazolidinediones
  Arms: Medical Therapy and Insulin Sensitizing (IS); Revascularization and Insulin Sensitizing (IS)
Drug: Insulin, sulfonylurea — Insulin, sulfonylurea
  Arms: Medical Therapy and Insulin Providing (IP); Revascularization and Insulin Providing (IP)
Drug: ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers — ACE Inhibitors, Angiotensin Receptor Blockers, Beta Blockers, Calcium Channel Blockers

SUMMARY:
The BARI 2D trial is a multicenter study that uses a 2x2 factorial design, with 2400 patients being assigned at random to initial elective revascularization with aggressive medical therapy or aggressive medical therapy alone with equal probability, and simultaneously being assigned at random to an insulin providing or insulin sensitizing strategy of glycemic control (with a target value for HbA1c of less than 7.0% for all patients).

SPECIFIC AIMS

A. Primary Aim

The primary aim of the BARI 2D trial is to test the following two hypotheses of treatment efficacy in 2400 patients with Type 2 diabetes mellitus and documented stable CAD, in the setting of uniform glycemic control and intensive management of all other risk factors including dyslipidemia, hypertension, smoking, and obesity:

1. Coronary Revascularization Hypothesis: a strategy of initial elective revascularization of choice (surgical or catheter-based) combined with aggressive medical therapy results in lower 5-year mortality compared to a strategy of aggressive medical therapy alone;
2. Method of Glycemic Control Hypothesis: with a target HbA1c level of less than 7.0%, a strategy of hyperglycemia management directed at insulin sensitization results in lower 5-year mortality compared to a strategy of insulin provision.

B. Secondary Aims

The secondary aims of the BARI 2D trial include: a) comparing the death, myocardial infarction or stroke combined endpoint event rate between the revascularization versus medical therapy groups and between the insulin sensitization versus insulin provision groups; b) comparing rates of myocardial infarction, other ischemic events, angina and quality of life associated with each revascularization and hyperglycemia management strategy; c) evaluating the relative economic costs associated with the trial treatment strategies, d) exploring the effect of glycemic control strategy on the progression and mechanism of vasculopathy including changes in PAI-1 gene expression.

DETAILED DESCRIPTION:
BACKGROUND:

Type 2 diabetes mellitus, which is becoming more prevalent in our society as the population ages, is one of the strongest risk factors for coronary artery disease (CAD) and consequent mortality. In addition to generating an enormous toll in human suffering, diabetes places an economic burden approaching 100 billion dollars annually on the U.S. health care system. Despite the well known dismal prognosis of diabetes complicated by angiographically documented CAD, the optimal treatment paradigm for this large group of patients has not been studied. Coronary revascularization, while increasingly used, has not been directly shown to be of additional benefit to simultaneous intensive medical management of CAD along with management of hyperglycemia, hypertension, dyslipidemia, and other risk factors. Moreover, while intensive efforts to lower HbA1c have been demonstrated to favorably affect the clinical course of Type 2 diabetes mellitus in terms of microvascular complications, the optimal hyperglycemia management strategy with regard to macrovascular outcome is not known.

These critical treatment dilemmas have motivated the development of BARI 2D, a multicenter randomized trial designed to determine in patients with Type 2 diabetes and stable CAD: 1) the efficacy of initial elective coronary revascularization combined with aggressive medical therapy, compared to an initial strategy of aggressive medical therapy alone; and 2) the efficacy of a strategy of providing more insulin (endogenous or exogenous), versus a strategy of increasing sensitivity to insulin (reducing insulin resistance), in the management of hyperglycemia, with a target HbA1c level of less than 7.0% for each strategy.

DESIGN NARRATIVE:

The BARI 2D trial is a multicenter study that uses a 2x2 factorial design, with 2400 patients being assigned at random to initial elective revascularization with aggressive medical therapy or aggressive medical therapy alone with equal probability, and simultaneously being assigned at random to an insulin providing or insulin sensitizing strategy of glycemic control (with a target value for HbA1c of less than 7.0% for all patients). Following confirmation of patient eligibility and provision of written consent, patients were randomized as shown below:

Number of Patients Per Treatment Assignment (N=2400 patients in total)

Stable Ischemic Heart Disease Treatment Strategy and Glycemic Control Strategy:

Revascularization and Insulin Providing (IP) N=600; Revascularization and Insulin Sensitizing (IS) N=600; Medical and Insulin Providing (IP) N=600; Medical and and Insulin Sensitizing (IS) N=600.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes mellitus
* Coronary arteriogram showing one or more vessels amenable to revascularization (greater than or equal to 50% stenosis)
* Objective documentation of ischemia OR subjectively documented typical angina with greater than or equal to 70% stenosis in at least one artery
* Suitability for coronary revascularization by at least one of the available methods (does not require the ability to achieve complete revascularization)
* Ability to perform all tasks related to glycemic control and risk factor management

Exclusion Criteria:

* Definite need for invasive intervention as determined by the attending cardiologist
* Prior bypass surgery (CABG) or prior catheter-based intervention within the 12 months before study entry
* Planned intervention for disease in bypass graft(s) if the patient is randomly assigned to a strategy of initial revascularization
* Class III or IV CHF
* Creatinine greater than 2.0 mg/dL
* HbA1c greater than 13%
* Need for major vascular surgery concomitant with revascularization (e.g., carotid endarterectomy)
* Left main stenosis greater than or equal to 50%
* Non-cardiac illness expected to limit survival
* Hepatic disease (ALT greater than 2 times the ULN)
* Fasting triglycerides greater than 1000 mg/dL in the presence of moderate glycemic control (HbA1c less than 9.0%)
* Current alcohol abuse
* Chronic steroid use judged to interfere with the control of diabetes, exceeding 10 mg of Prednisone per day or the equivalent
* Pregnancy, known, suspected, or planned in 5 years after study entry
* Geographically inaccessible or unable to return for follow-up
* Enrolled in a competing randomized trial or clinical study
* Unable to understand or cooperate with protocol requirements

Patients with Type 2 diabetes mellitus and CAD documented by coronary arteriography will be eligible for the trial if revascularization is not required for prompt control of severe or unstable angina. Diabetic patients who are being treated with insulin or oral hypoglycemic drugs will be eligible as well as diabetic patients treated with diet and exercise alone provided that a diagnosis of diabetes can be confirmed by record review or that a fasting plasma glucose (FPG) greater than 125/mg/dL (7.0 mmol/L) can be obtained. The determination of suitability for BARI 2D will be made by a physician-investigator at each participating institution on clinical grounds at the time of coronary angiography.

Significant CAD will be defined as at least one stenosis greater than 50%. Angina and ischemia will be assessed by use of patient self-report, physician examination, and appropriate diagnostic measures including exercise myocardial perfusion imaging, exercise echocardiography, exercise electrocardiography, and IV dipyridamole or adenosine myocardial perfusion imaging or invasively by doppler or pressure wire. Objective documentation of myocardial ischemia includes any of the following:

1. Exercise or pharmacologically-induced:

   1. Greater than or equal to 1 mm of horizontal or downsloping ST depression or elevation for greater than or equal to 60-80 milliseconds after the end of the QRS complex
   2. Myocardial perfusion defect
   3. Myocardial wall motion abnormality
2. Stabilized, prior acute coronary syndrome with CK-MB or troponin elevation or with new, greater than or equal to 0.5 mm ST depression or elevation, or T wave inversion of greater than or equal to 3 mm in 2 contiguous ECG leads
3. Doppler or pressure wire showing coronary flow reserve (CFR) less than 2.0 or fractional flow reserve (FFR) less than 0.75

Among patients without documented ischemia, only patients with stenosis greater than or equal to 70% presenting with classic anginal symptoms will be eligible for randomization.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2368 (Actual)
Dates: Start 2000-09; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chaitman, MD, Principal Investigator — St. Louis University; Robert L Frye, MD, Study Chair — Mayo Clinic; Mark Hlatky, Principal Investigator — Stanford University; Burton Sobel, Principal Investigator — University of Vermont & State Agricultural College; Sheryl F. Kelsey, PhD, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Background] Sobel BE, Frye R, Detre KM; Bypass Angioplasty Revascularization Investigation 2 Diabetes Trial. Burgeoning dilemmas in the management of diabetes and cardiovascular disease: rationale for the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial. Circulation. 2003 Feb 4;107(4):636-42. doi: 10.1161/01.cir.0000048897.03553.e4. PMID 12566379
- [Background] Brooks MM, Frye RL, Genuth S, Detre KM, Nesto R, Sobel BE, Kelsey SF, Orchard TJ; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial Investigators. Hypotheses, design, and methods for the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial. Am J Cardiol. 2006 Jun 19;97(12A):9G-19G. doi: 10.1016/j.amjcard.2006.02.023. Epub 2006 Apr 17. PMID 16813734
- [Background] Bypass Angioplasty Revascularization Investigation 2 Diabetes Study Group. Baseline characteristics of patients with diabetes and coronary artery disease enrolled in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Am Heart J. 2008 Sep;156(3):528-536, 536.e1-5. doi: 10.1016/j.ahj.2008.05.015. Epub 2008 Jul 31. PMID 18760137
- [Background] BARI 2D Study Group; Frye RL, August P, Brooks MM, Hardison RM, Kelsey SF, MacGregor JM, Orchard TJ, Chaitman BR, Genuth SM, Goldberg SH, Hlatky MA, Jones TL, Molitch ME, Nesto RW, Sako EY, Sobel BE. A randomized trial of therapies for type 2 diabetes and coronary artery disease. N Engl J Med. 2009 Jun 11;360(24):2503-15. doi: 10.1056/NEJMoa0805796. Epub 2009 Jun 7. PMID 19502645
- [Background] Brooks MM, Chung SC, Helmy T, Hillegass WB, Escobedo J, Melsop KA, Massaro EM, McBane RD, Hyde P, Hlatky MA; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Study Group. Health status after treatment for coronary artery disease and type 2 diabetes mellitus in the Bypass Angioplasty Revascularization Investigation 2 Diabetes trial. Circulation. 2010 Oct 26;122(17):1690-9. doi: 10.1161/CIRCULATIONAHA.109.912642. Epub 2010 Oct 11. PMID 20937978
- [Background] Grogan M, Jenkins M, Sansing VV, MacGregor J, Brooks MM, Julien-Williams P, Amendola A, Abbott JD; BARI 2D Study Group. Health insurance status and control of diabetes and coronary artery disease risk factors on enrollment into the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Diabetes Educ. 2010 Sep-Oct;36(5):774-83. doi: 10.1177/0145721710374653. Epub 2010 Jun 28. PMID 20584997
- [Background] Wall BM, Hardison RM, Molitch ME, Marroquin OC, McGill JB, August PA; BARI 2D Study Group. High prevalence and diversity of kidney dysfunction in patients with type 2 diabetes mellitus and coronary artery disease: the BARI 2D baseline data. Am J Med Sci. 2010 May;339(5):401-10. doi: 10.1097/MAJ.0b013e3181d430ad. PMID 20375690
- [Background] Rana JS, Hardison RM, Pop-Busui R, Brooks MM, Jones TL, Nesto RW, Bourassa MG; BARI 2D Investigators. Resting heart rate and metabolic syndrome in patients with diabetes and coronary artery disease in bypass angioplasty revascularization investigation 2 diabetes (BARI 2D) trial. Prev Cardiol. 2010 Summer;13(3):112-6. doi: 10.1111/j.1751-7141.2010.00067.x. PMID 20626665
- [Background] Thomas SB, Sansing VV, Davis A, Magee M, Massaro E, Srinivas VS, Helmy T, Desvigne-Nickens P, Brooks MM; BARI 2D Study Group. Racial differences in the association between self-rated health status and objective clinical measures among participants in the BARI 2D trial. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S269-76. doi: 10.2105/AJPH.2009.176180. Epub 2010 Feb 10. PMID 20147671
- [Background] Hlatky MA, Chung SC, Escobedo J, Hillegass WB, Melsop K, Rogers W, Brooks MM; BARI 2D Study Group. The effect of obesity on quality of life in patients with diabetes and coronary artery disease. Am Heart J. 2010 Feb;159(2):292-300. doi: 10.1016/j.ahj.2009.11.004. PMID 20152229
- [Background] Albu JB, Lu J, Mooradian AD, Krone RJ, Nesto RW, Porter MH, Rana JS, Rogers WJ, Sobel BE, Gottlieb SH; BARI 2D Study Group. Relationships of obesity and fat distribution with atherothrombotic risk factors: baseline results from the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Obesity (Silver Spring). 2010 May;18(5):1046-54. doi: 10.1038/oby.2009.339. Epub 2009 Oct 29. PMID 19875998
- [Background] Hlatky MA, Boothroyd DB, Melsop KA, Kennedy L, Rihal C, Rogers WJ, Venkitachalam L, Brooks MM; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Study Group. Economic outcomes of treatment strategies for type 2 diabetes mellitus and coronary artery disease in the Bypass Angioplasty Revascularization Investigation 2 Diabetes trial. Circulation. 2009 Dec 22;120(25):2550-8. doi: 10.1161/CIRCULATIONAHA.109.912709. Epub 2009 Nov 17. PMID 19920002
- [Background] Chaitman BR, Hardison RM, Adler D, Gebhart S, Grogan M, Ocampo S, Sopko G, Ramires JA, Schneider D, Frye RL; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Study Group. The Bypass Angioplasty Revascularization Investigation 2 Diabetes randomized trial of different treatment strategies in type 2 diabetes mellitus with stable ischemic heart disease: impact of treatment strategy on cardiac mortality and myocardial infarction. Circulation. 2009 Dec 22;120(25):2529-40. doi: 10.1161/CIRCULATIONAHA.109.913111. Epub 2009 Nov 17. PMID 19920001
- [Background] Kim LJ, King SB 3rd, Kent K, Brooks MM, Kip KE, Abbott JD, Jacobs AK, Rihal C, Hueb WA, Alderman E, Sing IR, Attubato MJ, Feit F; BARI 2D (Bypass Angioplasty Revascularization Investigation Type 2 Diabetes) Study Group. Factors related to the selection of surgical versus percutaneous revascularization in diabetic patients with multivessel coronary artery disease in the BARI 2D (Bypass Angioplasty Revascularization Investigation in Type 2 Diabetes) trial. JACC Cardiovasc Interv. 2009 May;2(5):384-92. doi: 10.1016/j.jcin.2009.01.009. PMID 19463459
- [Background] Schwartz L, Kip KE, Alderman E, Lu J, Bates ER, Srinivas V, Bach RG, Mighton LD, Feit F, King S 3rd, Frye RL; BARI 2D Study Group. Baseline coronary angiographic findings in the Bypass Angioplasty Revascularization Investigation 2 Diabetes trial (BARI 2D). Am J Cardiol. 2009 Mar 1;103(5):632-8. doi: 10.1016/j.amjcard.2008.11.024. Epub 2009 Jan 12. PMID 19231325
- [Background] Iskandrian AE, Heo J, Mehta D, Tauxe EL, Yester M, Hall MB, MacGregor JM. Gated SPECT perfusion imaging for the simultaneous assessment of myocardial perfusion and ventricular function in the BARI 2D trial: an initial report from the Nuclear Core Laboratory. J Nucl Cardiol. 2006 Jan-Feb;13(1):83-90. doi: 10.1016/j.nuclcard.2005.10.002. PMID 16464721
- [Background] Magee MF, Isley WL; BARI 2D Trial Investigators. Rationale, design, and methods for glycemic control in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial. Am J Cardiol. 2006 Jun 19;97(12A):20G-30G. doi: 10.1016/j.amjcard.2006.02.024. Epub 2006 Apr 19. PMID 16813735
- [Background] Barsness GW, Gersh BJ, Brooks MM, Frye RL; BARI 2D Trial Investigators. Rationale for the revascularization arm of the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial. Am J Cardiol. 2006 Jun 19;97(12A):31G-40G. doi: 10.1016/j.amjcard.2006.03.011. Epub 2006 Apr 17. PMID 16813736
- [Background] Sobel BE; BARI 2D Trial Investigators. Ancillary studies in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial: Synergies and opportunities. Am J Cardiol. 2006 Jun 19;97(12A):53G-58G. doi: 10.1016/j.amjcard.2006.03.013. Epub 2006 Apr 17. PMID 16813738
- [Background] Hlatky MA, Melsop KA, Boothroyd DB; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial Investigators. Economic evaluation of alternative strategies to treat patients with diabetes mellitus and coronary artery disease. Am J Cardiol. 2006 Jun 19;97(12A):59G-65G. doi: 10.1016/j.amjcard.2006.03.014. Epub 2006 Apr 7. PMID 16813739
- [Background] Escobedo J, Rana JS, Lombardero MS, Albert SG, Davis AM, Kennedy FP, Mooradian AD, Robertson DG, Srinivas VS, Gebhart SS; BARI 2D Study Group. Association between albuminuria and duration of diabetes and myocardial dysfunction and peripheral arterial disease among patients with stable coronary artery disease in the BARI 2D study. Mayo Clin Proc. 2010 Jan;85(1):41-6. doi: 10.4065/mcp.2009.0265. PMID 20042560
- [Background] McBane RD 2nd, Hardison RM, Sobel BE; BARI 2D Study Group. Comparison of plasminogen activator inhibitor-1, tissue type plasminogen activator antigen, fibrinogen, and D-dimer levels in various age decades in patients with type 2 diabetes mellitus and stable coronary artery disease (from the BARI 2D trial). Am J Cardiol. 2010 Jan 1;105(1):17-24. doi: 10.1016/j.amjcard.2009.08.643. Epub 2009 Nov 14. PMID 20102884
- [Background] Pop-Busui R, Lombardero M, Lavis V, Forker A, Green J, Korytkowski M, Sobel BE, Jones TL; BARI 2D Study Group. Relation of severe coronary artery narrowing to insulin or thiazolidinedione use in patients with type 2 diabetes mellitus (from the Bypass Angioplasty Revascularization Investigation 2 Diabetes Study). Am J Cardiol. 2009 Jul 1;104(1):52-8. doi: 10.1016/j.amjcard.2009.02.046. Epub 2009 May 13. PMID 19576321
- [Background] Schneider DJ, Hardison RM, Lopes N, Sobel BE, Brooks MM; Pro-Thrombosis Ancillary Study Group. Association between increased platelet P-selectin expression and obesity in patients with type 2 diabetes: a BARI 2D (Bypass Angioplasty Revascularization Investigation 2 Diabetes) substudy. Diabetes Care. 2009 May;32(5):944-9. doi: 10.2337/dc08-1308. Epub 2009 Feb 19. PMID 19228864
- [Background] Pop-Busui R, Lu J, Lopes N, Jones TL; BARI 2D Investigators. Prevalence of diabetic peripheral neuropathy and relation to glycemic control therapies at baseline in the BARI 2D cohort. J Peripher Nerv Syst. 2009 Mar;14(1):1-13. doi: 10.1111/j.1529-8027.2009.00200.x. PMID 19335534
- [Background] Pambianco G, Lombardero M, Bittner V, Forker A, Kennedy F, Krishnaswami A, Mooradian AD, Pop-Busui R, Rana JS, Rodriguez A, Steffes M, Orchard TJ. Control of lipids at baseline in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Prev Cardiol. 2009 Winter;12(1):9-18. doi: 10.1111/j.1751-7141.2008.00014.x. PMID 19301686
- [Background] Steiner G; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial Investigators. Statement of the problem. Am J Cardiol. 2006 Jun 19;97(12A):3G-8G. doi: 10.1016/j.amjcard.2006.02.022. Epub 2006 Apr 7. PMID 16813733
- [Background] Albu J, Gottlieb SH, August P, Nesto RW, Orchard TJ; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial Investigators. Modifications of coronary risk factors. Am J Cardiol. 2006 Jun 19;97(12A):41G-52G. doi: 10.1016/j.amjcard.2006.03.012. Epub 2006 Apr 19. PMID 16813737
- [Derived] Genuth SM, Vlachos H, Brooks MM, Bantle JP, Chaitman BR, Green J, Kelsey SF, King SB 3rd, McBane R, Sako EY, Schneider DJ, Steffes M, Frye RL; BARI 2D Study Group. BARI 2D: A Reanalysis Focusing on Cardiovascular Events. Mayo Clin Proc. 2019 Nov;94(11):2249-2262. doi: 10.1016/j.mayocp.2019.04.015. Epub 2019 Oct 4. PMID 31590967
- [Derived] Rezende PC, Everett BM, Brooks MM, Vlachos H, Orchard TJ, Frye RL, Bhatt DL, Hlatky MA. Hypoglycemia and Elevated Troponin in Patients With Diabetes and Coronary Artery Disease. J Am Coll Cardiol. 2018 Oct 9;72(15):1778-1786. doi: 10.1016/j.jacc.2018.07.067. PMID 30286920
- [Derived] Khan AA, Chung MJ, Novak E, Brown DL. Increased Hazard of Myocardial Infarction With Insulin-Provision Therapy in Actively Smoking Patients With Diabetes Mellitus and Stable Ischemic Heart Disease: The BARI 2D (Bypass Angioplasty Revascularization Investigation 2 Diabetes) Trial. J Am Heart Assoc. 2017 Sep 13;6(9):e005946. doi: 10.1161/JAHA.117.005946. PMID 28903941
- [Derived] Ikeno F, Brooks MM, Nakagawa K, Kim MK, Kaneda H, Mitsutake Y, Vlachos HA, Schwartz L, Frye RL, Kelsey SF, Waseda K, Hlatky MA; BARI-2D Study Group. SYNTAX Score and Long-Term Outcomes: The BARI-2D Trial. J Am Coll Cardiol. 2017 Jan 31;69(4):395-403. doi: 10.1016/j.jacc.2016.10.067. PMID 28126156
- [Derived] Wolk R, Bertolet M, Singh P, Brooks MM, Pratley RE, Frye RL, Mooradian AD, Rutter MK, Calvin AD, Chaitman BR, Somers VK; BARI 2D Study Group. Prognostic Value of Adipokines in Predicting Cardiovascular Outcome: Explaining the Obesity Paradox. Mayo Clin Proc. 2016 Jul;91(7):858-66. doi: 10.1016/j.mayocp.2016.03.020. Epub 2016 Jun 9. PMID 27289411
- [Derived] Damluji AA, Pomenti SF, Ramireddy A, Al-Damluji MS, Alfonso CE, Schob AH, Marso SP, Gilchrist IC, Moscucci M, Kandzari DE, Cohen MG. Influence of Total Coronary Occlusion on Clinical Outcomes (from the Bypass Angioplasty Revascularization Investigation 2 DiabetesTrial). Am J Cardiol. 2016 Apr 1;117(7):1031-8. doi: 10.1016/j.amjcard.2015.12.047. Epub 2016 Jan 14. PMID 26853953
- [Derived] Bittner V, Bertolet M, Barraza Felix R, Farkouh ME, Goldberg S, Ramanathan KB, Redmon JB, Sperling L, Rutter MK; BARI 2D Study Group. Comprehensive Cardiovascular Risk Factor Control Improves Survival: The BARI 2D Trial. J Am Coll Cardiol. 2015 Aug 18;66(7):765-773. doi: 10.1016/j.jacc.2015.06.019. PMID 26271057
- [Derived] Everett BM, Brooks MM, Vlachos HE, Chaitman BR, Frye RL, Bhatt DL; BARI 2D Study Group. Troponin and Cardiac Events in Stable Ischemic Heart Disease and Diabetes. N Engl J Med. 2015 Aug 13;373(7):610-20. doi: 10.1056/NEJMoa1415921. PMID 26267622
- [Derived] August P, Hardison RM, Hage FG, Marroquin OC, McGill JB, Rosenberg Y, Steffes M, Wall BM, Molitch M; BARI 2D Study Group. Change in albuminuria and eGFR following insulin sensitization therapy versus insulin provision therapy in the BARI 2D study. Clin J Am Soc Nephrol. 2014 Jan;9(1):64-71. doi: 10.2215/CJN.12281211. Epub 2013 Oct 31. PMID 24178969
- [Derived] Beohar N, Sansing VV, Davis AM, Srinivas VS, Helmy T, Althouse AD, Thomas SB, Brooks MM; BARI 2D Study Group. Race/ethnic disparities in risk factor control and survival in the bypass angioplasty revascularization investigation 2 diabetes (BARI 2D) trial. Am J Cardiol. 2013 Nov 1;112(9):1298-305. doi: 10.1016/j.amjcard.2013.05.071. Epub 2013 Aug 1. PMID 23910429
- [Derived] Bach RG, Brooks MM, Lombardero M, Genuth S, Donner TW, Garber A, Kennedy L, Monrad ES, Pop-Busui R, Kelsey SF, Frye RL; BARI 2D Investigators. Rosiglitazone and outcomes for patients with diabetes mellitus and coronary artery disease in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Circulation. 2013 Aug 20;128(8):785-94. doi: 10.1161/CIRCULATIONAHA.112.000678. Epub 2013 Jul 15. PMID 23857320
- [Derived] Pop-Busui R, Lu J, Brooks MM, Albert S, Althouse AD, Escobedo J, Green J, Palumbo P, Perkins BA, Whitehouse F, Jones TL; BARI 2D Study Group. Impact of glycemic control strategies on the progression of diabetic peripheral neuropathy in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Cohort. Diabetes Care. 2013 Oct;36(10):3208-15. doi: 10.2337/dc13-0012. Epub 2013 Jun 11. PMID 23757426
- [Derived] Althouse AD, Abbott JD, Sutton-Tyrrell K, Forker AD, Lombardero MS, Buitron LV, Pena-Sing I, Tardif JC, Brooks MM; BARI 2D Study Group. Favorable effects of insulin sensitizers pertinent to peripheral arterial disease in type 2 diabetes: results from the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Diabetes Care. 2013 Oct;36(10):3269-75. doi: 10.2337/dc12-2265. Epub 2013 Jun 4. PMID 23735723
- [Derived] Farkouh ME, Boden WE, Bittner V, Muratov V, Hartigan P, Ogdie M, Bertolet M, Mathewkutty S, Teo K, Maron DJ, Sethi SS, Domanski M, Frye RL, Fuster V. Risk factor control for coronary artery disease secondary prevention in large randomized trials. J Am Coll Cardiol. 2013 Apr 16;61(15):1607-15. doi: 10.1016/j.jacc.2013.01.044. PMID 23500281
- [Derived] Tamis-Holland JE, Lu J, Korytkowski M, Magee M, Rogers WJ, Lopes N, Mighton L, Jacobs AK; BARI 2D Study Group. Sex differences in presentation and outcome among patients with type 2 diabetes and coronary artery disease treated with contemporary medical therapy with or without prompt revascularization: a report from the BARI 2D Trial (Bypass Angioplasty Revascularization Investigation 2 Diabetes). J Am Coll Cardiol. 2013 Apr 30;61(17):1767-76. doi: 10.1016/j.jacc.2013.01.062. Epub 2013 Feb 28. PMID 23500245
- [Derived] Dagenais GR, Lu J, Faxon DP, Bogaty P, Adler D, Fuentes F, Escobedo J, Krishnaswami A, Slater J, Frye RL; BARI 2D Study Group. Prognostic impact of the presence and absence of angina on mortality and cardiovascular outcomes in patients with type 2 diabetes and stable coronary artery disease: results from the BARI 2D (Bypass Angioplasty Revascularization Investigation 2 Diabetes) trial. J Am Coll Cardiol. 2013 Feb 19;61(7):702-11. doi: 10.1016/j.jacc.2012.11.036. PMID 23410541
- [Derived] Brooks MM, Chaitman BR, Nesto RW, Hardison RM, Feit F, Gersh BJ, Krone RJ, Sako EY, Rogers WJ, Garber AJ, King SB 3rd, Davidson CJ, Ikeno F, Frye RL; BARI 2D Study Group. Clinical and angiographic risk stratification and differential impact on treatment outcomes in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Circulation. 2012 Oct 23;126(17):2115-24. doi: 10.1161/CIRCULATIONAHA.112.092973. Epub 2012 Sep 24. PMID 23008442
- [Derived] Schwartz L, Bertolet M, Feit F, Fuentes F, Sako EY, Toosi MS, Davidson CJ, Ikeno F, King SB 3rd. Impact of completeness of revascularization on long-term cardiovascular outcomes in patients with type 2 diabetes mellitus: results from the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D). Circ Cardiovasc Interv. 2012 Apr;5(2):166-73. doi: 10.1161/CIRCINTERVENTIONS.111.963512. Epub 2012 Apr 10. PMID 22496082
- [Derived] Cresci S, Wu J, Province MA, Spertus JA, Steffes M, McGill JB, Alderman EL, Brooks MM, Kelsey SF, Frye RL, Bach RG; BARI 2D Study Group. Peroxisome proliferator-activated receptor pathway gene polymorphism associated with extent of coronary artery disease in patients with type 2 diabetes in the bypass angioplasty revascularization investigation 2 diabetes trial. Circulation. 2011 Sep 27;124(13):1426-34. doi: 10.1161/CIRCULATIONAHA.111.029173. Epub 2011 Sep 12. PMID 21911782
- [Derived] Chung SC, Hlatky MA, Faxon D, Ramanathan K, Adler D, Mooradian A, Rihal C, Stone RA, Bromberger JT, Kelsey SF, Brooks MM; BARI 2D Study Group. The effect of age on clinical outcomes and health status BARI 2D (Bypass Angioplasty Revascularization Investigation in Type 2 Diabetes). J Am Coll Cardiol. 2011 Aug 16;58(8):810-9. doi: 10.1016/j.jacc.2011.05.020. PMID 21835316
- [Derived] Sobel BE, Hardison RM, Genuth S, Brooks MM, McBane RD 3rd, Schneider DJ, Pratley RE, Huber K, Wolk R, Krishnaswami A, Frye RL; BARI 2D Investigators. Profibrinolytic, antithrombotic, and antiinflammatory effects of an insulin-sensitizing strategy in patients in the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial. Circulation. 2011 Aug 9;124(6):695-703. doi: 10.1161/CIRCULATIONAHA.110.014860. Epub 2011 Jul 18. PMID 21768545
- [Derived] Chung SC, Hlatky MA, Stone RA, Rana JS, Escobedo J, Rogers WJ, Bromberger JT, Kelsey SF, Brooks MM. Body mass index and health status in the Bypass Angioplasty Revascularization Investigation 2 Diabetes Trial (BARI 2D). Am Heart J. 2011 Jul;162(1):184-92.e3. doi: 10.1016/j.ahj.2011.03.019. PMID 21742107
- [Derived] Beohar N, Davidson CJ, Massaro EM, Srinivas VS, Sansing VV, Zonszein J, Davis AM, Helmy T, Lopes NH, Thomas SB, Brooks MM. The impact of race/ethnicity on baseline characteristics and the burden of coronary atherosclerosis in the Bypass Angioplasty Revascularization Investigation 2 Diabetes trial. Am Heart J. 2011 Apr;161(4):755-63. doi: 10.1016/j.ahj.2010.12.013. PMID 21473976
- [Derived] Dagenais GR, Lu J, Faxon DP, Kent K, Lago RM, Lezama C, Hueb W, Weiss M, Slater J, Frye RL; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Study Group. Effects of optimal medical treatment with or without coronary revascularization on angina and subsequent revascularizations in patients with type 2 diabetes mellitus and stable ischemic heart disease. Circulation. 2011 Apr 12;123(14):1492-500. doi: 10.1161/CIRCULATIONAHA.110.978247. Epub 2011 Mar 28. PMID 21444887
- See also: Click here for the BARI 2D Study Web site — http://www.bari2d.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2,368 patients were enrolled at 49 clinical centers from United States, Canada, Brazil, Mexico, Czech Republic, and Austria between January 1, 2001 and March 31, 2005. Each of the 2368 patients was simultaneously assigned to initial revascularization or medical therapy and assigned to insulin providing or insulin sensitizing therapy.
Period: Overall Study
Arm/Group | Revascularization and Insulin Providing (IP) | Revascularization and Insulin Sensitizing (IS) | Medical Therapy and Insulin Providing (IP) | Medical Therapy and Insulin Sensitizing (IS)
Started | 592 | 584 | 593 | 599
Completed | 575 | 574 | 578 | 585
Not Completed | 17 | 10 | 15 | 14
Not completed — Withdrawal by Subject | 17 | 10 | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revascularization and Insulin Providing (IP) | Revascularization and Insulin Sensitizing (IS) | Medical Therapy and Insulin Providing (IP) | Medical Therapy and Insulin Sensitizing (IS) | Total
Number analyzed (Participants) | 592 | 584 | 593 | 599 | 2368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 362 | 354 | 350 | 373 | 1439
  >=65 years | 230 | 230 | 243 | 226 | 929
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.5) | 62.4 (9.1) | 62.7 (8.8) | 62.2 (9.3) | 62.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 172 | 172 | 182 | 702
  Male | 416 | 412 | 421 | 417 | 1666
Region of Enrollment [Number; unit: participants]
  United States | 376 | 367 | 376 | 380 | 1499
  Canada | 87 | 88 | 89 | 89 | 353
  Brazil | 89 | 89 | 89 | 89 | 356
  Mexico | 21 | 21 | 22 | 21 | 85
  Europe | 19 | 19 | 17 | 20 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality
Time Frame: five years
Population: Intention to treat analysis (ITT) of the two main effects in the 2x2 factorial design, 1) Revascularization versus Medical Therapy and 2) Insulin Sensitizing (IS) versus Insulin Providing (IP)
Measure: Number; unit: participants
Arm/Group | Revascularization and Insulin Providing (IP) | Revascularization and Insulin Sensitizing (IS) | Medical Therapy and Insulin Providing (IP) | Medical Therapy and Insulin Sensitizing (IS)
Number analyzed (Participants) | 592 | 584 | 593 | 599
participants | 80 | 75 | 80 | 81
Statistical Analysis 1: Comparison: Revascularization and Insulin Providing (IP) vs Revascularization and Insulin Sensitizing (IS) vs Medical Therapy and Insulin Providing (IP) vs Medical Therapy and Insulin Sensitizing (IS); Test type: Superiority or Other; p = 0.97, Log Rank — A separate test with alpha=0.05 was conducted for each treatment comparison of the main effects in the 2x2 factorial design; Risk Difference (RD) = -0.005, 95% CI 2-sided [-0.031 to 0.020] — Risk difference of all-cause mortality for Revascularization compared with Medical therapy
Statistical Analysis 2: Comparison: Revascularization and Insulin Providing (IP) vs Revascularization and Insulin Sensitizing (IS) vs Medical Therapy and Insulin Providing (IP) vs Medical Therapy and Insulin Sensitizing (IS); Test type: Superiority or Other; p = 0.89, Log Rank — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.003, 95% CI 2-sided [-0.029 to 0.022] — Risk difference of all-cause mortality for Insulin Sensitizing glycemic control strategy compared with Insulin Providing glycemic control strategy

2. Secondary Outcome: Number of Participants With Death, Myocardial Infarction, or Stroke
Time Frame: five years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Revascularization and Insulin Providing (IP) | Revascularization and Insulin Sensitizing (IS) | Medical Therapy and Insulin Providing (IP) | Medical Therapy and Insulin Sensitizing (IS)
Number analyzed (Participants) | 592 | 584 | 593 | 599
participants | 145 | 121 | 143 | 140
Statistical Analysis 1: Comparison: Revascularization and Insulin Providing (IP) vs Revascularization and Insulin Sensitizing (IS) vs Medical Therapy and Insulin Providing (IP) vs Medical Therapy and Insulin Sensitizing (IS); Test type: Superiority or Other; p = 0.70, Log Rank — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.013, 95% CI 2-sided [-0.049 to 0.022] — Risk difference of Death/MI/Stroke for Revascularization compared with Medical Therapy
Statistical Analysis 2: Comparison: Revascularization and Insulin Providing (IP) vs Revascularization and Insulin Sensitizing (IS) vs Medical Therapy and Insulin Providing (IP) vs Medical Therapy and Insulin Sensitizing (IS); Test type: Superiority or Other; p = 0.13, Log Rank — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.024, 95% CI [-0.060 to 0.012] — Risk difference of Death/MI/Stroke for Insulin Sensitizing glycemic control strategy compared with Insulin Providing glycemic control strategy

ADVERSE EVENTS:
Time Frame: 5 years
Description: Clinic visits conducted monthly for first 6 months and every 3 months thereafter until the study ended.
Arm/Group | Revascularization and Insulin Providing (IP) | Revascularization and Insulin Sensitizing (IS) | Medical Therapy and Insulin Providing (IP) | Medical Therapy and Insulin Sensitizing (IS)
Serious Adverse Events (participants affected / at risk) | 230/592 | 210/584 | 230/593 | 235/599
Other Adverse Events (participants affected / at risk) | 331/592 | 362/584 | 344/593 | 363/599
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revascularization and Insulin Providing (IP) (N=592) | Revascularization and Insulin Sensitizing (IS) (N=584) | Medical Therapy and Insulin Providing (IP) (N=593) | Medical Therapy and Insulin Sensitizing (IS) (N=599)
Death (Cardiac disorders) | 80 | 75 | 80 | 81
Myocardial Infarction (Cardiac disorders) | 67 | 51 | 71 | 67
Stroke (Vascular disorders) | 17 | 13 | 19 | 14
Severe Hypoglycemia (Endocrine disorders) | 46 | 36 | 62 | 32
Congestive Heart Failure (Cardiac disorders) | 111 | 119 | 107 | 129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revascularization and Insulin Providing (IP) (N=592) | Revascularization and Insulin Sensitizing (IS) (N=584) | Medical Therapy and Insulin Providing (IP) (N=593) | Medical Therapy and Insulin Sensitizing (IS) (N=599)
Pitting Edema (General disorders) | 293 | 317 | 304 | 335
Bone Fracture (Musculoskeletal and connective tissue disorders) | 38 | 48 | 36 | 34
Laser Therapy for Macular Edema (Eye disorders) | 47 | 42 | 52 | 54
Lower Extremity Ulcer (Vascular disorders) | 55 | 55 | 48 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No